CLINICAL TRIAL: NCT01752829
Title: A Single-arm, Observational, Post-marketing Study to Evaluate the Effects of the A.M.I. Protector Adjustable Gastric Band on Weight Loss, Co-morbidities, Adverse Events and Other Clinical Characteristics.
Brief Title: Post-marketing Surveillance Study of A.M.I. Protector Adjustable Gastric Band
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Weight to Go Ltd (Other)
Responsible Party: Sponsor
Other Study IDs: Version PBS.V2.11.12
Record Dates: First submitted 2012-12-11; First posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Obesity
Keywords: Obesity; gastric; banding; Weight; co-morbidities; dilatation; Excess weight loss; adjustable gastric banding
MeSH Terms: conditions — Obesity; Body Weight; Dilatation, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The laparoscopic adjustable gastric band (LAGB) is a safe and effective surgical intervention for chronically obese patients who have exhausted all non-surgical weight loss treatments. Numerous published studies have confirmed both the safety and efficacy of the LAGB and its beneficial impact on obesity-associated conditions, such as type 2 diabetes, joint and back pain and hypertension. The A.M.I. Protector Band is a modification of an existing gastric band (the A.M.I. Soft Gastric Band) which has been in use since 2001 and which has been shown to be both safe and effective. The specific design modification is in the form of a section of mesh, which provides support to the gastric pouch and which further restricts food portion sizes. The expectation is that this will deliver optimal weight loss whilst having the maximum possible impact on obesity-associated conditions such as type 2 diabetes and hypertension. In the longer term, there is also the possibility that the Protector Band will reduce the incidence of band complications such as slippage and dilatation (or stretching) of the gastric pouch. In this study we will recruit approximately 200 patients who will then undergo surgical implantation of the A.M.I. Protector Band. The study participants will then be followed for a period of 3-years, during which time we will record weight loss, changes in co-morbid conditions such as diabetes and the incidence of band complications, including slippage and pouch dilatation.

DETAILED DESCRIPTION:
Where patients express an interest in the A.M.I. Protector Band, they will be given a Patient Information Sheet which will form the basis of a discussion with the attending physician. Patients opting for the Protector Band will be told that their anonymised clinical data will be stored in a secure database and used for research purposes. They will also be required to attend for regular follow-up (see below) for a period of three years after implantation.

Following this initial consultation, a minimum period of 2-weeks will be required before the patient is listed for surgery. This will provide a suitable period during which the patient can consider the options and seek clarification on any points about which they are unclear.

In the case of the A.M.I. Protector Band the surgery will be performed in two locations:

* Spire Hospital Parkway (Birmingham)
* Spire Hospital Manchester

All band procedures will be performed by one of two surgeons; Mr. Paul Super and Prof. Franco Favretti according to a standard protocol.

In all cases, informed consent will be obtained prior to surgery.

Patients will remain in hospital overnight and be discharged the following day.

On discharge, patients will be given comprehensive written instructions regarding optimal nutritional and physical activity. They will also be provided with a 24-hour, Emergency Helpline number in the event of problems.

All patients will be followed for a period of three years, with a formal review at 5 weeks and then at 3, 6, 9, 12, 18, 24 and 36 months. However, patients will be free to attend additional clinics between the formal reviews should they wish. At each visit the patient's weight, height, waist/hip ratio and blood pressure (BP) will be recorded. In addition, a range of blood tests will be carried out at baseline, at 12, 24 and 36 months. A self-administered Quality of Life questionnaire will be completed prior to surgery and then at 12, 24 and 36 months of follow-up.

At the completion of the 3-year study, patients will be able to transition into our usual care gastric band programme for long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* obese subjects with BMI >30kg/m2 with one or more co-morbidities
* Obese subjects with BMI >40kg/m2 with or without co-morbidities

Exclusion Criteria:

* previous history of drug abuse
* history of bleeding disorders
* On long-term steroid therapy
* Pregnancy
* Previous gastric surgery
* Chronic lung disease
* history of psychotic disease
* Inflammatory bowel disease
* Unstable angina or dysrhythmia
* liver cirrhosis
* Autoimmune disease (SLE etc)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese subjects who are candidates for gastric banding
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Percentage excess weight loss (%EWL) | 3 years

SECONDARY OUTCOMES:
Impact of weight loss on co-morbidities such as type 2 diabetes, hypertension etc | 3-years
Incidence of band-related complications such as band slippage; erosion; port/tubing complications; port/band infection; pouch dilatation | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr David Ashton, MD PhD, Principal Investigator — Weight to Go Ltd
Locations (1):
- Weight To Go Ltd, Birmingham, United Kingdom